CLINICAL TRIAL: NCT04136405
Title: Cross Sectional Survey on the Burden, Impacts and Causes of Hepatitis C Virus (HCV) Outbreak in South West Region in Burkina Faso
Acronym: REVERSO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Centre Muraz (Other); Université Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: ANRS 12389 REVERSO
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Hepatitis C Virus Infection, Past or Present; Chronic Hepatitis c
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates hepatitis C virus (HCV) outbreak in South West general population in Burkina Faso with three specific objectives: estimate HCV prevalence in South West Region general population in 2019; identify factors associated with recent HCV infection (in subjects younger than 20 years); and evaluate the pilot treatment strategy implemented by the national program for diagnosed cases during investigation.

DETAILED DESCRIPTION:
A previous ANRS (French National Agency for Research on AIDS and Viral Hepatitis)12270 study supported by Burkina Faso's Minister of Health, used blood samples from the 2010 Demographic and Health Survey (DHS) to document the country's national and regional prevalences and highlighted a localized HCV epidemic in the Southwest Region with a prevalence of 13.2% which was 4 times higher than the national prevalence. This high prevalence of HCV was found in both adults and youth.

Given the particular epidemiological situation of the South-West region and the limits of the 2010 DHS, we aimed to carry out a thorough investigation of this HCV epidemic in the South-West region of Burkina Faso in order to control it.

A mixed methodology (quantitative and qualitative) will be used including: (i) a cross-sectional survey to estimate the prevalence of HCV infection in the South-West population in Burkina Faso; (ii) a case-control study among individuals less than 20 years of age to identify factors associated with current HCV transmission; (iii) a qualitative survey to provide additional information explaining the high prevalence of HCV infection (historical events, for example); (iv) a cohort study to evaluate a pilot treatment management strategy to be implemented by the national program in the South West Region

ELIGIBILITY:
Inclusion Criteria:

* To be a usual resident of the Burkina Faso South West region
* Express informed consent

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: General population of South West region of Burkina Faso
Sampling Method: Probability Sample
Enrollment: 3300 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
HCV seroprevalence | at inclusion (cross-sectional survey)
  proportion of individuals with a past or present HCV infection (rapid test)

SECONDARY OUTCOMES:
Chronic hepatitis C prevalence | at inclusion (cross-sectional survey)
  proportion of individuals with chronic hepatitis (plasma HCV viral load by PCR)

CONTACTS AND LOCATIONS:
Locations (1):
- Région du Sud-Ouest, Gaoua, Burkina Faso